CLINICAL TRIAL: NCT05170347
Title: Ocular Graft-Versus-Host-Disease After Allogeneic Haematopoietic Stem Cell Transplantation: A Territory-Wide Prospective Cohort
Brief Title: oGVHD After Bone Marrow Transplantation: a Territory-wide Cohort
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Allie Lee, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 21-145
Record Dates: First submitted 2021-06-11; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Graft Vs Host Disease; Haematological Malignancy; Cancer
Keywords: Graft Vs Host Disease; Bone Marrow Transplant; Cancer; Haematological malignancy
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Conjunctival samples will be stored for further investigation of ocular microbiome in laboratory.
  Blood and tear samples will be stored for detection of biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-Haematopoietic Stem Cell Transplantation (Post-HSCT) patients: * Patient aged 18 or above
  * Underwent allogeneic HSCT in Queen Mary Hospital(QMH) in the two-year recruitment period
- Family Control Subjects: The research team will invite an accompanying family member to be the family control. Microbiome and tear samples will be collected for comparison. The sample collection schedule is the same as the corresponding post-HSCT case.

SUMMARY:
Allogeneic Haematopoietic stem cell transplantation (HSCT) is an effective treatment for all array of blood or blood-producing organ disorders. Graft-versus-host-disease (GVHD) occurs as a result of an overactive immunological system against normal host tissues. It can happen in the liver, skin, mucosal surface of the eye, gastrointestinal tract, and genitalia.

Ocular GVHD occurs in 30-70% of patients after HSCT. It mainly affects the ocular surface, including the conjunctiva and cornea. In severe cases, multiple clinical manifestations can lead to painful non-healing corneal ulcers, secondary infections, and visual loss.

oGVHD can be debilitating and severely impact patients' quality of life. However, there are no widely accepted guidelines available for prevention and management.

In collaboration with the Department of Haematology of Queen Mary Hospital, the investigators set out to establish a territory-wide cohort of patients receiving HSCT. Primarily, the investigators aim to establish the population-based epidemiology of oGVHD and understand the natural history and the long-term ophthalmic outcomes of oGVHD via this study.

DETAILED DESCRIPTION:
Allogeneic haematopoietic stem cell transplantation (HSCT) is an effective treatment for all array of haematological disorders. Graft-versus-host-disease (GVHD) occurs as a result of an overactive systemic immunological response against normal host tissues, in particular the liver, skin, mucosal surface of the eye, gastrointestinal tract, and genitalia.

Ocular graft-versus-host-disease (oGVHD) occurs in 30-70% patients after allogeneic HSCT. It mainly affects the ocular surface, and pathologically it is characterized by decreased conjunctival goblet cell density, increased conjunctival squamous metaplasia, and infiltration of tissues with inflammatory cells. Common clinical manifestations include keratoconjunctivitis sicca, marginal keratitis, conjunctivitis, and conjunctival scarring, and anterior uveitis. In severe cases, these can lead to painful non-healing corneal ulcers, secondary infections, and visual loss. Risk factors for oGVHD reported in the literature included non- Caucasian race, male recipient from female donor, more extensive and severe systemic involvement, pre-existing diabetes mellitus, and use of anti-thymocyte globulin.

oGVHD can be debilitating and severely impact patients' quality of life. Although common and significant, currently there are no widely accepted guidelines available for prophylaxis and management.

The Haemopoietic Stem Cell Transplantation Centre at Queen Mary Hospital is the only quaternary referral centre for adults in Hong Kong since 1990 and now it serves over 100 patients per year. In collaboration with the Department of Haematology of QMH, the investigators set out to establish a territory-wide cohort of patients receiving allogeneic HSCT to fill the current knowledge gaps.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or above
* Underwent allogeneic HSCT in QMH in the two-year recruitment period

Exclusion Criteria:

* Underwent autologous HSCT
* Patient unable to attend follow-up visits

Family Control Subjects The research team will invite an accompanying family member to be the family control. Microbiome and tear samples will be collected for comparison. The sample collection schedule is the same as the corresponding post-HSCT case.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In a two-year recruitment period, all patients attending the pre-HSCT assessment clinic in the Bone Marrow Transplant Centre (BMTC) at Queen Mary Hospital (QMH) will be invited to join the cohort. The sample size is estimated to be 250. This is based on the calculation that, each year, approximately 120-130 patients underwent allogeneic HSCT at the BMTC of QMH.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Population-based epidemiology of oGVHD after allogeneic HSCT | 5 years, starting from the baseline visit
  Incidence of oGVHD at 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, and 60 months following allogeneic HSCT (according to ? criteria)

SECONDARY OUTCOMES:
Longitudinal change in OSDI scores | 5 years, starting from the baseline visit
  Change in OSDI scores post-BMT over the 5-year study period will be evaluated. OSDI scores are calculated from a Chinese-validated OSDI questionnaire. They assess oGVHD-induced dry eye disease symptom severity and their burden on the patients' quality of life.
Serial changes in the anatomy, function & quantity of Meibomian gland | 5 years, starting from the baseline visit
  Since Meibomian gland dysfunction is one of the main clinical features of oGVHD, anatomical, functional and quantitative changes of Meibomian gland will be examined. Parameters associated with Meibomian gland anatomy and quantity include its level of obstruction and dropout, which can be observed from Meibographs taken with the Keratography 5M and LipiView devices. With the help of the ImageJ software, these parameters will be graded according to the () criteria. Degree of Meibomian gland atrophy indicates the functionality of the Meibomian gland thus the degree of Meibomian gland dysfunction.
Prevalence of ocular surface disease pre-BMT | 5 years, starting from the baseline visit
  (Purpose). The presence of ocular surface disease will be confirmed through a comprehensive eye examination (visual acuity, intraocular pressure, slit-lamp and fundus examination), Pentacam, specular microscopy (corneal cell density), and tear assessment (tear breakup time (TBUT), fluorescein staining pattern, non-anaesthetic Schirmer's test).
Compositional and density changes in ocular surface microbiome over time | 5 years, starting from the baseline visit
  Changes in diversity and density of microbial colonies on the ocular surface are hypothesised to be involved in oGVHD pathogenesis, and hence are investigated.
Proteomics of tear secretions | 5 years, starting from the baseline visit
  oGVHD is an ocular complication arisen from the infiltration of inflammatory cells. The presence, type and quantity of inflammatory markers implied in oGVHD pathogenesis will be confirmed through proteomic analysis. Tear matrix metalloproteinase-9 (MMP-9) will be the main inflammatory marker investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Allie Lee, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Ophthalmology, LKS Faculty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arai S, Jagasia M, Storer B, Chai X, Pidala J, Cutler C, Arora M, Weisdorf DJ, Flowers ME, Martin PJ, Palmer J, Jacobsohn D, Pavletic SZ, Vogelsang GB, Lee SJ. Global and organ-specific chronic graft-versus-host disease severity according to the 2005 NIH Consensus Criteria. Blood. 2011 Oct 13;118(15):4242-9. doi: 10.1182/blood-2011-03-344390. Epub 2011 Jul 26. PMID 21791424
- [Background] Zeiser R, Blazar BR. Pathophysiology of Chronic Graft-versus-Host Disease and Therapeutic Targets. N Engl J Med. 2017 Dec 28;377(26):2565-2579. doi: 10.1056/NEJMra1703472. No abstract available. PMID 29281578
- [Background] Aronni S, Cortes M, Sacchetti M, Lambiase A, Micera A, Sgrulletta R, Bonini S. Upregulation of ICAM-1 expression in the conjunctiva of patients with chronic graft-versus-host disease. Eur J Ophthalmol. 2006 Jan-Feb;16(1):17-23. doi: 10.1177/112067210601600104. PMID 16496240
- [Background] Kim SK. Ocular graft vs. host disease. Ocul Surf. 2005 Oct;3(4 Suppl):S177-9. doi: 10.1016/s1542-0124(12)70250-1. PMID 17216114
- [Background] Wang JC, Teichman JC, Mustafa M, O'Donnell H, Broady R, Yeung SN. Risk factors for the development of ocular graft-versus-host disease (GVHD) dry eye syndrome in patients with chronic GVHD. Br J Ophthalmol. 2015 Nov;99(11):1514-8. doi: 10.1136/bjophthalmol-2014-306438. Epub 2015 May 6. PMID 25947556
- [Background] Ogawa Y, Kim SK, Dana R, Clayton J, Jain S, Rosenblatt MI, Perez VL, Shikari H, Riemens A, Tsubota K. International Chronic Ocular Graft-vs-Host-Disease (GVHD) Consensus Group: proposed diagnostic criteria for chronic GVHD (Part I). Sci Rep. 2013 Dec 5;3:3419. doi: 10.1038/srep03419. PMID 24305504
- [Background] Na KS, Yoo YS, Mok JW, Lee JW, Joo CK. Incidence and risk factors for ocular GVHD after allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2015 Nov;50(11):1459-64. doi: 10.1038/bmt.2015.187. Epub 2015 Aug 24. PMID 26301966
- [Background] Tabbara KF, Al-Ghamdi A, Al-Mohareb F, Ayas M, Chaudhri N, Al-Sharif F, Al-Zahrani H, Mohammed SY, Nassar A, Aljurf M. Ocular findings after allogeneic hematopoietic stem cell transplantation. Ophthalmology. 2009 Sep;116(9):1624-9. doi: 10.1016/j.ophtha.2009.04.054. PMID 19729097
- See also: Adult HSCT, Hong Kong West Cluster, Hospital Authority, Hong Kong — https://www3.ha.org.hk/hkwc/transplantservice/HSCT-Adult.html

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT05170347/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT05170347/ICF_001.pdf